CLINICAL TRIAL: NCT03154281
Title: A Phase 1 Evaluation of the Safety and Tolerability of Niraparib in Combination With Everolimus in Advanced Gynecologic Malignancies and Breast Cancer
Brief Title: Evaluation of the Safety and Tolerability of Niraparib With Everolimus in Advanced Gynecologic Malignancies and Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNE001
Record Dates: First submitted 2017-05-08; First posted 2017-05-16 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Breast; Ovarian
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — niraparib; Everolimus

STUDY DESIGN:
Intervention Model Description: The statistical analysis will be mainly descriptive. Continuous variables will be summarized using descriptive statistics: N, mean, standard deviation, median, minimum and maximum. Categorical variables will be presented using frequencies and percentages. Time-to-event will be described by N, median, range, number censored, and Kaplan-Meier plots. A traditional dose escalation design will be used, beginning with the lowest dose level and escalating to the maximum allowable dose level as specified in the protocol. Three patients will be treated one at a time at a given dose level. A maximum of 4 dosing levels results in a maximum sample size of n=24 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): (each cycle is 28 days long) Everolimus 5mg daily on Mondays, Wednesdays, and Fridays Niraparib 100mg daily
  Interventions: Drug: niraparib; Drug: everolimus
- Cohort 2 (Experimental): (each cycle is 28 days long) Everolimus 5 mg daily on Mondays, Wednesdays, and Fridays Niraparib 200 mg daily
  Interventions: Drug: niraparib; Drug: everolimus
- Cohort 3 (Experimental): (each cycle is 28 days long) Everolimus 5 mg daily Niraparib 200 mg daily
  Interventions: Drug: niraparib; Drug: everolimus
- Cohort 4 (Experimental): (each cycle is 28 days long) Everolimus 5 mg daily Niraparib 300 mg daily
  Interventions: Drug: niraparib; Drug: everolimus

INTERVENTIONS:
Drug: niraparib — Niraparib 100 mg will be administered orally once daily continuously. Niraparib will be administered as a flat-fixed dose (100mg, 200 mg, or 300 mg daily) depending on the cohort the patient is enrolled to, and not by body weight or body surface area. Each dose should be swallowed whole without chewing. The consumption of water is permissible. Patients should take doses at approximately the same times each day, and record this information in the patient diary. Patients will be provided with a diary in which to record their intake of study drug. However, the actual number of doses taken by the patient must be calculated from the number of tablets dispensed and returned.
  Other Names: MK-4827
Drug: everolimus — Everolimus 5 mg tablets will be used. Everolimus will be self-administered orally on a daily basis and doses will either be 5 mg (1 tablet) thrice weekly or 5 mg daily depending on the cohort the patient is enrolled to. Each cycle will be 28 days; everolimus will be taken continuously with no rest between cycles.
  Other Names: Afinitor

SUMMARY:
Open-label, cohort study to determine the feasibility and tolerability of the combination of daily niraparib and daily or thrice weekly everolimus for one 28-day cycle in patients with advanced ovarian and breast cancer.

DETAILED DESCRIPTION:
The goal of this study is to determine a maximum tolerated dose of the combination of niraparib and everolimus. To do this, investigators will estimate the maximum tolerated dose that is defined as the dose level at which less than one-third of patients will experience a dose-limiting toxicity. A traditional dose escalation design will be used, beginning with the lowest dose level and escalating to the maximum allowable dose level as specified in the protocol. One of the following outcomes will determine the treatment of subsequent patients:

* If none of the three patients experiences a dose-limiting toxicity , the next group of patients will be entered in the next higher dose cohort. All patients within a cohort must have completed at least one cycle (28 days) prior to initiation of the next cohort of patients.
* If one of the three patients experiences a dose-limiting toxicity , three more patients will be accrued at the current dose level. Subsequently, if only one of the six patients treated at this level experiences a dose-limiting toxicity , the dose will be escalated to the next higher dose in the next group of patients. If two or more of the six patients experiences a dose-limiting toxicity , the maximum tolerated dose has been exceeded and is defined as the previous dose at which no more than 1/3 experienced a dose-limiting toxicity .
* If at least two of the three experience a dose-limiting toxicity , the maximum tolerated dose has been exceeded and is defined as the previous dose at which no more than 1/3 experienced a dose-limiting toxicity .

If the lowest allowable dose level exceeds the maximum tolerated dose, the study will be terminated and the combination will not be deemed safe for use in this population. Additionally, the highest dose level will not be exceeded, even if no dose-limiting toxicities are experienced at that dose.

Investigators will summarize the adverse events overall and by individual adverse event categories. Serious adverse events will be summarized in a similar manner. These summaries will be performed overall and for each dose cohort. Investigators will summarize all events as well as the highest grade for a given subject. Investigators will summarize the number of subjects that exhibit a dose-limiting toxicity at each dose cohort and describe the dose-limiting toxicity for each subject, if applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a gynecologic malignancy or breast cancer (triple negative or hormone receptor positive only) that is refractory/intolerant to all therapies known to confer clinical benefit in the advanced or metastatic setting or if the patient's clinical team and the PI believe that the study treatment gives the patient the best chance for clinical benefit
2. Patients with breast cancer must have measurable disease per RECIST 1.1. criteria. Patients with ovarian cancer are eligible with or without measurable disease
3. Patients with ovarian cancer must have had appropriate surgical management for their disease and should be platinum resistant (recurrence within 6 months of last platinum-containing regimen) or be refractory to platinum-containing regimens
4. Patients with endometrial, cervical, or any other advanced gynecologic malignancy must have already received or not be a candidate for all therapy proven to have a survival benefit
5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
6. Patients must be ≥18 years of age
7. Patients must have adequate organ function, defined as follows:

   * Absolute neutrophil count ≥1,500/µL
   * Platelets ≥125,000/µL
   * Hemoglobin ≥10 g/dL
   * Serum creatinine ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation
   * Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤1 x ULN
   * Aspartate aminotransferase and alanine aminotransferase ≤2.5 x ULN unless liver metastases are present, in which case they must be ≤5 x ULN
8. Patient agrees to blood draws during screening and at the end of treatment for molecular and cytogenetic analysis
9. Female patients of childbearing potential must have a negative serum pregnancy test (beta hCG) at Screening
10. Female patients of childbearing potential must agree to use an acceptable method of birth control (excluding hormonal birth control methods, see Section 3.0.5) for 72 hours prior to initiation of therapy and to continue its use during the study and for at least 180 days after the final dose
11. Male patients must agree to use an acceptable form of birth control (see Section 3.0.5) from study Day 1 through at least 180 days after the final dose
12. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Patients with HER2+ breast cancer measured by standard IHC or FISH testing
2. Patients must not be simultaneously enrolled in any other interventional clinical trial
3. Patients must not have had major surgery ≤3 weeks of starting the study and patient must have recovered from any effects of any major surgery
4. Patients must not have had investigational therapy administered ≤4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study
5. Patients must not have had radiotherapy encompassing >20% of the bone marrow
6. Patients must not have received prior treatment with a known PARP inhibitor or have participated in a study where any treatment arm included administration of a known PARP inhibitor
7. Patients must not have a known hypersensitivity to the components of niraparib, everolimus, rapamycin analogues, or the excipients
8. Patients must not be immunocompromised (patients with splenectomy are allowed)
9. Patients must not have had any known, persistent >Grade 2 toxicity from prior cancer therapy
10. Patients must not have had any known, persistent (>4 weeks), ≥Grade 3 hematological toxicity or fatigue from prior cancer therapy
11. Patients must not have received a transfusion (platelets or red blood cells) ≤4 weeks of the first dose of study treatment
12. Patients must not have current evidence of any condition, therapy, or laboratory abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study or interfere with the patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate
13. Patients must not have had diagnosis, detection, or treatment of another type of cancer ≤2 years prior to randomization (except basal or squamous cell carcinoma of the skin that has been definitively treated)
14. Patients must not have known, symptomatic brain or leptomeningeal metastases
15. Patients must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, interstitial lung disease, HIV or Hepatitis B, or any psychiatric disorder that prohibits obtaining informed consent
16. Patients must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
17. Patient is a woman with a positive serum pregnancy test ≤3 days prior to study drug administration, is breast-feeding, or is planning to conceive children within the projected duration of the study treatment
18. Patients with uncontrolled or poorly controlled hypertension
19. Patients taking ACE inhibitors (patients that have no known medical reason to require therapy with ACE inhibitors may be switched to another appropriate antihypertensive treatment prior to initiation of study treatment)
20. Patients taking strong or moderate CYP3A4/PgP inhibitors or strong CYP3A4/PgP inducers (appendix 2) (if medically appropriate, patients may be switched to another appropriate therapy at least 14 days prior to initiation of study treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Williams, Principal Investigator — Avera Cancer Institute
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at Avera Cancer Institute in Sioux Falls, South Dakota, United States from July 2017 to May 2021.
Pre-assignment Details: A total of 14 participants with a gynecologic malignancy or breast cancer (triple negative or hormone receptor positive only) were enrolled in this study.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 8 | 6 | 0 | 0
Completed | 7 | 4 | 0 | 0
Not Completed | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dose limiting toxicity (DLT) was observed in 2 patients in Cohort 2. Patients were not enrolled in higher dose Cohorts per study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 8 | 6 | 0 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 3 | 4 |  |  | 7
  >=65 years | 5 | 2 |  |  | 7
Age, Continuous [Median (Full Range); unit: years] | 67.5 [51 to 71] | 62 [51 to 77] |  |  | 64.5 [51 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 |  |  | 14
  Male | 0 | 0 |  |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 |  |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Does-limiting Toxicity (DLT)
Description: The DLT criteria for adverse events occurring in Cycle 1 while determining the maximum tolerated dose (MTD) are described in the protocol. The number of patients who experience DLT from the trial treatment is recorded.
Time Frame: From the start of treatment to 30 days after the first dose of study drug
Population: No patient was enrolled in Cohort 3 or Cohort 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 6 | 0 | 0
Participants | 0 | 2 | 0 | 0

2. Secondary Outcome: Number of Patients With Beneficial Clinical Response
Description: Tumor objective response is evaluated according to RECIST 1.1 response criteria. Number of patients with beneficial clinical response (SD, PR and CR) are recorded in each group.
Time Frame: From beginning of study to the end of the 2nd cycle, and then at 16 weeks if the patient has stable disease or better.
Population: One out of eight patients in Cohort 1 was not evaluable due to rapid progression in cycle 1.
  One out of six patients in Cohort 2 was not evaluable due to DLT and treatment was discontinued in cycle 1.
  No patients was enrolled in Cohort 3 or Cohort 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 5 | 0 | 0
Participants | 5 | 2 | 0 | 0

3. Secondary Outcome: Number of Patients With Tumor Objective Response
Description: Tumor objective response is evaluated according to RECIST 1.1 response criteria. Number of patients with beneficial clinical response (PR and CR) are recorded in each group.
Time Frame: From beginning of study to the end of the 2nd cycle, and then at 16 weeks if the patient has stable disease or better.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 5 | 0 | 0
Participants | 2 | 0 | 0 | 0

4. Other Pre Specified Outcome: Progression Free Survival (in Months)
Description: Tumor assessment according to RECIST 1.1 was performed at the end of the second cycle, and then again at 16 weeks if the patient has stable disease or better. Scans may be performed every 8-12 weeks thereafter at the discretion of the investigators.
Time Frame: From beginning of study to the end of the 2nd cycle, and then at 16 weeks if the patient has stable disease or better
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 5 | 0 | 0
months | 3.7 [1.2 to 7.3] | 2.4 [1.8 to 6.8] |  |

5. Other Pre Specified Outcome: Overall Survival
Description: Survival status was monitored every 8 weeks for 2 years following the last dose
Time Frame: From the end of treatment till 2 years following the last dose
Population: No patients were enrolled in Cohort 3 or Cohort 4 Two patients in Cohort 1 were alive at the end of follow up at 2 years after the last dose.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 6 | 0 | 0
months | 16.1 [1.9 to 36.4] | 16.6 [4.3 to 32.5] |  |

ADVERSE EVENTS:
Time Frame: From beginning of treatment to 30 days after the last dose. The duration for collecting adverse events ranges from 2 months to 1 year, depending on the length of study treatment for each patient.
Description: no patients was enrolled in cohort 3 or cohort 4
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/8 | 5/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=6) | Cohort 3 (N=0) | Cohort 4 (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=6) | Cohort 3 (N=0) | Cohort 4 (N=0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (6) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (7) | 4 (8) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (7) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 3 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 3 (7) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 5 (11) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT03154281/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03154281/ICF_001.pdf